CLINICAL TRIAL: NCT02639130
Title: Quantification of the Contribution of GLP-1 to Mediating Insulinotropic Effects of DPP-4 Inhibition With Vildagliptin in Healthy Subjects and Type 2-diabetic Patients Using Exendin [9-39] as a GLP-1 Receptor Antagonist
Brief Title: GLP-1 Mediating DPP-4 Inhibition in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diabeteszentrum Bad Lauterberg im Harz (Other)
Responsible Party: Principal Investigator, Michael A. Nauck, Prof. Dr. med. Michael A. Nauck, Diabeteszentrum Bad Lauterberg im Harz
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DZBL-2007-1
Record Dates: First submitted 2015-12-17; First posted 2015-12-24 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
Keywords: Gastric Inhibitory Polypeptide (GIP); Glucagon-Like Peptide 1 (GLP-1); DPP-4 inhibition; Exendin [9-39]; Gastric emptying; Glucagon; Incretin; Insulin Secretion; Normal glucose-tolerant
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vildagliptin (Active Comparator): After a screening examination, patients were treated with vildagliptin and participated in meal tests (day 9 and 10, respectively), in a crossover design. Between the two treatment periods, there was a ≥ 5 week wash-out period.
  Experimental procedures: Meal test, determination of the rate of gastric emptying. On days 9 and 10 of treatment, the volunteers underwent a mixed meal (one scrambled egg, a slice of ham, 10 g of butter, two slices of toast, 20 g strawberry jam, and 200 ml of unsweetened tea) test in the morning after fasting overnight. 13C-octanoic acid (110 µl/100 mg) was used as label.
  Meal tests were performed (days 9 and 10), without and with a high dose intravenous infusion of exendin [9-39].
  Interventions: Drug: Exendin [9-39]; Drug: Placebo
- Placebo (Placebo Comparator): After a screening examination, patients were treated with placebo, and participated in meal tests (day 9 and 10, respectively), in a crossover design. Between the two treatment periods, there was a ≥ 5 week wash-out period.
  Experimental procedures: Meal test, determination of the rate of gastric emptying. On days 9 and 10 of treatment, the volunteers underwent a mixed meal (one scrambled egg, a slice of ham, 10 g of butter, two slices of toast, 20 g strawberry jam, and 200 ml of unsweetened tea) test in the morning after fasting overnight. 13C-octanoic acid (110 µl/100 mg) was used as label.
  Meal tests were performed (days 9 and 10), without and with a high dose intravenous infusion of exendin [9-39].
  Interventions: Drug: Exendin [9-39]; Drug: Placebo

INTERVENTIONS:
Drug: Exendin [9-39] — Exendin [9-39] at 350 and 500 pmol/kg/min for infusion as challenge agent
  Other Names: (GLP-1 receptor antagonist)
Drug: Placebo — Placebo infusion as challenge agent

SUMMARY:
To determine the extent to which the effects of treatment with LAF237 100 mg QD on glucagon secretion are mediated by Glucagon-like-peptide 1 (GLP-1) in type 2 diabetic patients and healthy subjects.

DETAILED DESCRIPTION:
Design:

This two center study employs a double blind, placebo controlled, cross-over study in patients with type 2 diabetes (T2D) and healthy volunteers with comparable age, gender and BMI distribution. Subjects (40 patients and 40 healthy volunteers, referred to as subjects in remaining part of the document) will be randomized to 100 mg LAF 237 QD or placebo for two 10-day treatment periods in a cross-over design. Thirty two (32) efficacy evaluable patients are required to complete the study.

Each subjects will participate in an approximate 14-day screening period, a 2-week wash-out period from metformin, a 1-day baseline period and a 10-day treatment period followed by a 2-4 week wash-out period and a second treatment period. An end of study evaluation will be conducted following the completion of the second treatment period or in the event of early withdrawal or termination of the patient.

At screening, subjects meeting inclusion/exclusion criteria will begin a weight maintenance diet containing 50% carbohydrates, 30% protein and 20% fat. Patients will receive guidance on dietary maintenance at screening and will stay on this diet from screening to the end of study evaluation. Following the screening visit, enrolled patients will start a 2 week drug wash-out period where oral hypoglycemic medication will be discontinued.

During the drug wash-out period, all patients will monitor their glucose levels two times a day (prior to breakfast and dinner) using a glucometer. Additionally, at one week intervals, patients will perform a seven point blood glucose test, where glucose measurements will be made prior to and two hours after each meal, and prior to bed. Weekly telephone calls will be made to each patient, where the results of these glucose tests will be recorded. Patients will be discontinued from the study during the wash-out period if fasting glucose levels exceed 200 mg/dl on any two consecutive measurements.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with either diet/exercise or metformin
* HbA1c 6.5 - 9.0 %
* Fasting plasma glucose 6.0 - 11.0 mmol/l
* Body-mass-index 20.0 - 35.0 kg/m²
* Healthy controls were required to have a normal oral glucose tolerance test (75g) and no first-degree relatives with type 2 diabetes nor a personal history of gestational diabetes

Exclusion Criteria:

* Significant heart, kidney (serum creatinine ≤ 123 µmol/l in woman and ≤ 132 µmol/l in men), liver (transaminases < 2fold upper limit of normal) and gastrointestinal disease

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Ratio of integrated insulin secretion rates (total AUC ISR) over 4 hour following the meal | 4 hour following the meal
total AUC Glucose over 4 hour following the meal | 4 hour following the meal

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Nauck, Prof., Principal Investigator — Diabeteszentrum Bad Lauterberg
Locations (1):
- Diabeteszentrum Bad Lauterberg, Bad Lauterberg im Harz, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nauck MA, Kind J, Kothe LD, Holst JJ, Deacon CF, Broschag M, He YL, Kjems L, Foley J. Quantification of the Contribution of GLP-1 to Mediating Insulinotropic Effects of DPP-4 Inhibition With Vildagliptin in Healthy Subjects and Patients With Type 2 Diabetes Using Exendin [9-39] as a GLP-1 Receptor Antagonist. Diabetes. 2016 Aug;65(8):2440-7. doi: 10.2337/db16-0107. Epub 2016 Apr 5. PMID 27207543